CLINICAL TRIAL: NCT05227170
Title: Impact of Lp299v on Vascular Function in Patients With PASC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Professor of Medicine and Pharmacology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRO42931
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: endothelial function; PASC; COVID-19; inflammation; microbiome
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lp299v (Experimental): Subjects will consume 20 billion colony forming units of Lp299v (2 capsules) once daily for 8 weeks.
  Interventions: Other: Lactobacillus Plantarum 299v Freeze Dried Capsule
- Heat-killed placebo control (Placebo Comparator): Subjects will consume potato starch (2 capsules) once daily for 8 weeks.
  Interventions: Other: Freeze Dried Potato Starch Capsule

INTERVENTIONS:
Other: Lactobacillus Plantarum 299v Freeze Dried Capsule — The intervention is a probiotic lactobacillus that is contained in food products in the US
  Arms: Lp299v
Other: Freeze Dried Potato Starch Capsule — The intervention is potato starch that is freeze dried designed to mimic the lp299v capsule.
  Arms: Heat-killed placebo control

SUMMARY:
Emerging data show that SARS-CoV-2 infection causes gut microbiome changes strongly associated with Post-Acute Sequelae of SARS-CoV-2 (PASC). The investigators and others have established that an orally ingested probiotic (Lactobacillus plantarum 299v, Lp299v) reduces circulating levels of cell-free mitochondrial DNA (cf-mtDNA), decreases toll-like receptor 9 (TLR9) activation [and downstream interleukin (IL-6)], and improves micro- and macrovascular (brachial artery) endothelial dysfunction [as measured by flow-mediated dilation (FMD%)] in humans. Recently published data also report impaired brachial FMD% and increased vascular stiffness post-SARS-CoV-2 infection. Based on these data, the investigators hypothesize that supplementation with Lp299v will attenuate SARS-CoV-2 associated endothelial dysfunction by reducing cf-mtDNA, TLR9 activation, and inflammation.

DETAILED DESCRIPTION:
The intestinal immune system plays a critical role in systemic immunity, and its interaction with the systemic immune system plays a crucial role in determining the severity and outcomes of common pulmonary infections. SARS-CoV-2 infection alters the composition and metabolism of the gut microbiome. Greater losses of beneficial species in the human gut microbiome of SARS-CoV-2 patients are associated with severe disease and greater systemic inflammation. These pathological alterations are observed at least 6 months post-infection and are associated with greater residual systemic inflammation and PASC symptoms.

Six weeks of Lp299v supplementation in otherwise healthy smokers reduces circulating levels of the pro-inflammatory IL-6 and reduces monocyte adhesion to endothelial cells. IL-6 is elevated in patients with PASC and strongly correlates with TLR9 activation in disease states with high circulating cf-mtDNA levels. We published trial data showing once daily Lp299v supplementation (20 billion colony forming units/day) in men with coronary artery disease (CAD) improves endothelium-dependent vasodilation in the brachial artery and NO-dependent vasodilation of resistance arterioles from CAD patients. Further, preliminary data suggest Lp299v reduces circulating levels of cf-mtDNA (Fig. 2B). We also published data showing that 6 weeks of Lp299v has a significant anti-inflammatory effect on PBMC gene transcription, with gene ontology analyses indicating Lp299v supplementation inhibits TLR9 activation (z-score -3.48, P<0.0000000023). Combining the evidence that Lp299v reduces (1) circulating cf-mtDNA; (2) TLR9 activation; and (3) IL-6 levels while improving micro- and macrovascular endothelial function make Lp299v an excellent candidate to test as an intervention to improve vascular function in PASC patients.

Therefore, we will recruit subjects ages ≥18-89 who carry a clinical diagnosis of PASC and are within a window of 30-180-day post-acute symptom resolution into an 8-week, double-blind, randomized, placebo-controlled clinical trial of Lp299v supplementation. Measurements of micro- and macrovascular function, systemic inflammation, and stool microbiota composition will be made.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 89 years
* 30-180 days post-COVID-19 diagnosis
* PASC diagnosed based on symptom report/expert physician judgement

Exclusion Criteria:

* Antibiotics within four weeks of enrollment
* History of chronic diseases (renal insufficiency, liver dysfunction, cancer requiring systemic treatment within 3 years of enrollment)
* History of cognitive impairment/inability to follow study procedures
* Short gut syndrome, inflammatory bowel disease, or an ileostomy.
* Subjects currently taking Vitamin K antagonists such as coumadin or warfarin
* Pregnant at the time of screening
* Unstable coronary artery disease (new symptoms or event within 30 days of enrollment)
* Daily alcohol use (may interfere with Lp299v's action)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow Mediated Dilation (FMD%) | 8 weeks
  This is a measurement of endothelial function in the brachial artery

SECONDARY OUTCOMES:
Nitroglycerin-Mediated Vasodilation of the brachial artery (NMD) | 8 weeks
  Measurement of vascular smooth muscle reactivity
Hyperemic Flow Velocity | 8 weeks
  Measurement of microvascular endothelial function
Carotid-Femoral Pulse Wave Velocity (cfPWV) | 8 weeks
  Measurement of vascular stiffness
Percentage of Laser Doppler Signal | 8 weeks
  Measurement of skin microvascular function
interleukin-6 | 8 weeks
  circulating inflammatory marker
Stool microbiota alpha diversity | 8 weeks
  Diversity of bacterial species in the individual microbiome
Stool microbiota beta diversity | 8 weeks
  Differences in bacterial composition between intervention arms
Cell-Free Mitochondrial DNA (cf-mtDNA) | 8 weeks
  Level of circulating cf-mtDNA in the plasma
Brachial Artery Resting Diameter | 8 weeks
  resting diameter of the brachial artery - representative of resting vascular tone
Myeloid Cell Population phenotypes | 8 weeks
  Quantification and identification of mononuclear cell and neutrophil types

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Within 1 year of completion of all studies procedures.